CLINICAL TRIAL: NCT01755910
Title: Effect of Thoracic Paravertebral Block on the Autonomous System as Measured by Heart Rate Variability (HRV)
Brief Title: Effect of Thoracic Paravertebral Block on Heart Rate Variability (HRV)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Marina Simaioforidou, Anesthesiologist, Larissa University Hospital
Other Study IDs: HRV Thoracic paravertebral
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Breast Surgery; Thoracic Paravertebral Block; HRV; Autonomic Nervous System
Keywords: Breast Surgery; Thoracic Paravertebral Block; HRV; Autonomic Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left thoaracic paravertebral block: Surgery in the left breast under left thoracic paravertebral block and HRV
  Interventions: Other: Left thoracic paravertebral block
- Right thoracic paravertebral block and HRV: Surgery in the right breast under right thoracic paravertebral block and HRV
  Interventions: Other: Right thoracic paravertebral block

INTERVENTIONS:
Other: Left thoracic paravertebral block
  Groups: Left thoaracic paravertebral block
Other: Right thoracic paravertebral block
  Groups: Right thoracic paravertebral block and HRV

SUMMARY:
The Left thoracic paravertebral block have a different effect on heart's autonomic nervous system, as measured with Heart Rate Variability, compared to Right interscalene block

ELIGIBILITY:
Inclusion Criteria:

* Elective breast surgery
* Age 20 - 65 years
* ASA I - II

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the thoracic paravertebral block
* Severe kyphoscoliosis
* Allergy to local anesthetics
* BMI > 35
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication
* Arrythmia
* Ischaemic heart disease
* Diabetes mellitus
* Thyroid function disorders
* Patients with conduction disorders on the ECG
* Electrolyte disorders (K+, Na+, Ca++)
* Patients on medication that affect the ECG

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for elective breast surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Effect of thoracic paravertebral block on Heart Rate Variability (HRV) | 30 min after the application of the thoracic paravertebral block
  The Left thoracic paravertebral block has different effect on heart's autonomic nervous system, as measured with HRV, than the Right.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Simaioforidou, Medicine, Principal Investigator — Larissa University Hospital; George Vretzakis, Medicine, Study Director — Larissa University Hospital; Aikaterini Tsiaka, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Larissa University Hospital, Larissa, Thessally, Greece